CLINICAL TRIAL: NCT04735471
Title: A Phase 1 Safety and Efficacy Study of ADI-001 Anti-CD20 CAR-engineered Allogeneic Gamma Delta (γδ) T Cells in Adults With B Cell Malignancies
Brief Title: A Phase 1 Study of ADI-001 in B Cell Malignancies
Acronym: GLEAN-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated - Halted Prematurely
Sponsor: Adicet Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADI-20200101
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma, Follicular; Lymphoma, Mantle-Cell; Marginal Zone Lymphoma; Primary Mediastinal B-cell Lymphoma; Diffuse Large B Cell Lymphoma; Lymphoma, Non-Hodgkin
Keywords: B-cell lymphoma; CAR-T; Cell Therapy; Allogeneic Cell Therapy; T cells, gamma delta; Immunotherapy, Adoptive; Antigens, CD20
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ADI-001 Dose Escalation (Experimental): ADI-001 is administered via infusion with ascending dose levels as a single dose to determine the maximum tolerated dose (MTD) or maximum assessed dose (MAD) of ADI-001 (Part 1a).
  Interventions: Genetic: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- ADI-001 Dose Extension (Experimental): ADI-001 is administered via infusion at MAD/MTD to evaluate the safety of multiple doses (Part 1b).
  Interventions: Genetic: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- ADI-001 Dose Expansion (Experimental): Dose Expansion ADI-001 is administered via infusion at the MTD/MAD to confirm recommended phase 2 dose (Part 2).
  Interventions: Genetic: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ADI-001 — Anti-CD20 CAR-T
Drug: Fludarabine — Chemotherapy for Lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for Lymphodepletion

SUMMARY:
This is a Phase 1 dose escalation study following a 3+3 study design. The purpose of this study is to evaluate the safety and efficacy of ADI-001 in patients with B cell malignancies.

DETAILED DESCRIPTION:
ADI-001 is an investigational immunotherapy composed of allogeneic gamma delta T cells that is being evaluated as a potential treatment for patients diagnosed with B cell malignancies who have relapsed or are refractory to at least two prior regimens. This first-in-human study will assess the safety and tolerability of ADI-001 and is designed to determine the maximum tolerated dose (MTD) or maximum assessed dose (MAD). Patients will be administered a single infusion or multiple infusions of ADI-001 cells. The study will include the following two parts:

Part 1 : dose escalation and extension. Parts 1a (escalation) and 1b (extension) will involve escalation and administration of single dose of ADI-001 and multiple doses of ADI-001.

Part 2 : dose expansion will involve dose administration of ADI-001 at MTD/MAD as determined in Part 1.

The study will also assess the pharmacokinetics and pharmacodynamics of ADI-001.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory (R/R) previously treated B cell malignancies.
2. Prior treatment must include at least 2 prior regimens, including anti CD20 antibody therapies. Prior Treatment with CD19 CAR T may be considered.
3. Documented measurable disease as defined by Lugano 2014
4. Male or female ≥ 18 years of age
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
6. Adequate hematological, renal, pulmonary, cardiac, and liver function
7. Female patients who are not pregnant or breastfeeding
8. Female patients of childbearing potential and all male patients must agree to use highly effective methods of birth control for the duration of the study.

Exclusion Criteria:

1. Current or history of any of the following conditions:

   1. Central nervous system (CNS) primary lymphoma (current or history)
   2. Unrelated malignancy requiring systemic treatment (current or history [in the past 3 years, other than hormonal treatment which is allowed])
2. Any of the following current conditions:

   1. Active acute or chronic graft versus host disease (GvHD) other than grade 1 with skin involvement, or GvHD requiring immunosuppressive treatment within 4 weeks of enrollment
   2. Any other acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration
   3. Tumor mass effects such as bowel obstruction or blood vessel compression that require therapy
   4. Opportunistic infections
3. History of any clinically significant conditions in the opinion of the Investigator
4. Prior treatment with any of the following:

   a Gene therapy, genetically modified cell therapy, or adoptive T cell therapy within 6 weeks of study enrollment.

   b Radiation therapy within 4 weeks prior to study entry. Palliative local radiation may be allowed within 1 week prior to study entry.

   c Autologous stem cell transplant (SCT) within 6 weeks of planned ADI 001 infusion.

   d Allogeneic transplant and donor lymphocyte infusion within 3 months of planned CAR T cell infusion
5. Patients unwilling to participate in an extended safety monitoring period (long term follow up [LTFU] protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
The Incidence of Subjects with Dose Limiting Toxicities within each dose level cohort | Day 28
  This primary endpoint will be used to determine the Maximum Tolerated Dose (MTD) or Maximum Assessed dose (MAD).
Proportion of treatment emergent and treatment related adverse events | 1 year
  This primary endpoint will be used to determine the MTD/MAD of ADI-001

SECONDARY OUTCOMES:
Frequency and persistence of ADI-001 | Day 1 through Month 12
  Defined as duration from Day 1 to undetectable levels of ADI-001 cells per microliter blood
Overall Response Rate by Lugano Criteria | Day 28, Month 3, 6, 9, and 12
Duration of Response | Day 28, Month 3, 6, 9, and 12
Progression Free Survival | Day 28, Month 3, 6, 9, and 12
Time To Progression | Day 28, Month 3, 6, 9, and 12
Overall Survival | Day 28, Month 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Adicet Medical Director, Study Director — Adicet Bio
Locations (10):
- United States (10):
  - Stanford University Medical Center, Stanford, California
  - University of Miami- Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northside Hospital Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - The State University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Roswell Park Cancer Institute, Buffalo, New York
  - Baylor Scott & White Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nishimoto KP, Barca T, Azameera A, Makkouk A, Romero JM, Bai L, Brodey MM, Kennedy-Wilde J, Shao H, Papaioannou S, Doan A, Masri C, Hoang NT, Tessman H, Ramanathan VD, Giner-Rubio A, Delfino F, Sharma K, Bray K, Hoopes M, Satpayev D, Sengupta R, Herrman M, Abbot SE, Aftab BT, An Z, Panuganti S, Hayes SM. Allogeneic CD20-targeted gammadelta T cells exhibit innate and adaptive antitumor activities in preclinical B-cell lymphoma models. Clin Transl Immunology. 2022 Feb 2;11(2):e1373. doi: 10.1002/cti2.1373. eCollection 2022. PMID 35136603